CLINICAL TRIAL: NCT06071481
Title: Efficacy, Safety and Dose Response of Vitamin D in Prevention of Dengue Haemorrhagic Fever and Dengue Shock Syndrome- A Phase 2 Open-label Randomized Controlled Trial
Brief Title: Role of Vitamin D in Prevention of Dengue Haemorrhagic Fever and Dengue Shock Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Fazle Rabbi Chowdhury, Associate Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2023/4579
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue | interventions — JPT1 protein, human; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Arm-1: Standard treatment, Arm-2: Standard treatment and 2,00,000 IU Vitamin D oral solution, Arm 3: Standard treatment and 4,00,000 IU Vitamin D oral solution
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm-1 (No Intervention): Standard supportive care ( Plenty of oral fluid, Tab. Paracetamol 500mg)
- Arm-2 (Experimental): Standard supportive treatment + 2,00,000 IU Vitamin D oral solution
  Interventions: Drug: Arm-2 : 2,00,000 IU Vitamin D3 oral solution , Arm-3: 4,00,000 IU Vitamin D3 oral solution
- Arm-3 (Experimental): Standard supportive treatment + 4,00,000 IU Vitamin D oral solution
  Interventions: Drug: Arm-2 : 2,00,000 IU Vitamin D3 oral solution , Arm-3: 4,00,000 IU Vitamin D3 oral solution

INTERVENTIONS:
Drug: Arm-2 : 2,00,000 IU Vitamin D3 oral solution , Arm-3: 4,00,000 IU Vitamin D3 oral solution — 2,00,000 IU Vitamin D3 oral solution in the form of cholecalciferol 4,00,000 IU Vitamin D3 oral solution in the form of cholecalciferol
  Arms: Arm-2; Arm-3

SUMMARY:
Dengue is an arthropod-borne disease, found in tropical and sub-tropical climates worldwide, mostly in urban and semi-urban areas. Unfortunately, there is no intervention available to stop dengue severity. Despite significant efforts into developing vaccine and antiviral drug for dengue fever over the years, numerous challenges remain before an efficient, safe vaccine and antiviral drug. Dengue Haemorrhagic Fever (DHF) and Dengue Shock Syndrome (DSS) are a serious form of dengue infection that can escalate in a non-negligible percentage of febrile patients. Factors responsible for this deterioration are weakly understood. The host's genetics and secondary infections from novel dengue serotypes are obvious risk factors. The dietary state of the host has also been emphasized as a potentially important predictor of progression because some nutrients have potent immunomodulatory effects. Vitamin D is particularly important as it has ability to control immunological processes, including the downregulation of pro-inflammatory Th1 activity, which has been linked to the pathophysiology of severe dengue. There is a preliminary study regarding the effectiveness of vitamin D in the prevention of DHF and DSS in human. But a larger study is needed to prove its utility. The objective of the study is to determine the role of Vitamin D in efficacy, safety and dose response in the prevention of DHF and DSS. This will be an open-label Phase-2 Randomized controlled trial (RCT) which will be carried out in Dengue cell, Emergency Department and Outpatient Department (OPD) of Medicine Department in Bangabandhu Sheikh Mujib Medical University, Dhaka. It will be conducted from September 2023 to August 2024 enrolling about 120 patients from Dengue cell, Emergency Department and OPD of Medicine Department BSMMU. The duration of the study will be one year. All the investigations will be done in BSMMU. Patients will be followed up by phone call and physical visit. Those with severe symptoms will be admitted and evaluated accordingly. The study will have three arms namely, Arm 1(receiving standard care), Arm 2(receiving standard care and 2,00,000 IU Vitamin D oral solution) and Arm 3(receiving standard treatment and 4,00,000 IU Vitamin D oral solution). The patients will be enrolled according to inclusion criteria (having age more than 18 to 65years, NS1 positive, fever more than ≥38°C for 3days or less, typical sign symptoms of Dengue fever) and exclusion criteria (>72hours of fever, critically ill patients, pregnancy, known Vitamin D hypersensitivity, high serum calcium level, hypoalbuminaemia, malignancy, known nephrolithiasis and severe renal impairment). Information will be obtained on socio-demographic and clinical characteristics through face to face interview using a structured questionnaire. Clinical data and relevant blood samples will be taken at first appointment then after 4th day and 8th day of enrollment. This study has minimal chance of physical risks. Study purpose will be explained to the participants and informed written consent will be taken before collection of data. Data will be collected with assurance of proper safety and privacy. The interventional drug, vitamin D3 is a widely used agent with rare minimal side effects like, vomiting, abdominal pain, headache, constipation etc. Each participant will be counselled about the outcome of the drug and will be followed up and managed for potential side effects. Participants will be identified by a code number, strict confidentiality and anonymity will be maintained. There will be no loss of work time and no compensation will be available for the participants as this will be a part of standard care. On the other hand, this study would be helpful for both the clinician and the patients in making a rational approach in Group A Dengue fever for the prevention of DHF and DSS. Prior to the commencement of this study, the research protocol will take approval from Research and Training Monitoring Department(RTMD) of BCPS. The analyzed data will be presented in the form of text, tables, and graphs. Finally collected data will be analyzed by graph pad prism. Statistical analysis will be performed by Chi-square test on categorical data and one way ANOVA with Tukey's multiple comparisons test on continuous data. Kaplan-Meier Curve will be used to study the progression into DHF and DSS. This study, for the first time in Bangladesh, will obtain the baseline data regarding the utility of Vitamin D therapy in Dengue uncomplicated cases in preventing further deterioration of clinical severity and mortality. This trial will help clinicians and policy makers to avail a possible repurposing of Vitamin D for prevention of severe dengue. In addition, it will guide designing larger study to generate strong evidence and change the national health response accordingly.

DETAILED DESCRIPTION:
Rationale of the Study: Bangladesh is a hyperendemic region for dengue infection and is inflicted with massive outbreaks throughout nations since 2019. According to DGHS report, the highest admissions due to dengue infection was recorded in 2019. Last year, in 2022 total number of death was 281, which was the highest in terms of mortality since 2000. It is disturbing to notice that, this year up to August 11th, 2023 the number of mortality reached 373, which has already exceeded the previous records. Most of our population is exposed to dengue infection and it is proven that secondary infection with a different serotype likely manifests as severe form of dengue. This may be the very reason for unprecedented rise in mortality, as antibody dependent enhancement in secondary dengue with memory T cell response are central to development of severe dengue infections. Proinflammatory cytokines released from T cell and macrophages along with complement breakdown products are found to be the main offender in DHF and DSS that increases vascular permeability of endothelium and organ dysfunction. Unfortunately, there is no antiviral agent that has been proven to work in dengue infection and vaccination is not an option in Bangladesh so we can only provide supportive treatment and observe until warning signs appear. After deterioration we admit the patient for more agile monitoring and give intravenous fluids as required and in negligible cases, steroids and other organ support. Researchers are now trying to target this cytokine storm and finding a way to reverse this effect in initial days of dengue infection. So a new intervention is needed to halt this disease progression. There is however emerging evidence of role of nutrients in immunomodulation. Vitamin D is a promising agent proved by preliminary studies. In those previous studies vitamin D showed potential as an immunomodulatory agent that may have a role in controlling dengue severity by downregulation of pro-inflammatory Th1 activity and reduction of the surface expression of C- type lectin, specially "mannose receptor" which is the known primary receptor for DENV attachment on macrophages that trigger immune signalling and rapid rise in cytokine production. There is only one human RCT that has concluded a possible role of this agent. Keeping all the evidences in mind this trial is designed to prove the efficacy, safety and dose response of vitamin D in the prevention of dengue severity and mortality. This study may aid in proving a strong empirical evidence base to support the role of vitamin D in reducing admission and thereby mortality. In addition, it will guide designing larger study to generate strong evidence and change the national health response accordingly.

Research question:

Is vitamin D effective and safe in the prevention of progression to DHF and DSS?

Objectives:

General Objectives:

To determine the efficacy, safety and dose response of Vitamin D in prevention of DHF and DSS.

Specific Objectives:

1. To find out the efficacy of Vitamin D in reducing dengue mortality and describe the percentage reduction.
2. To find out the safety of using Vitamin D in dengue fever and delineate it's safety profile.
3. To compare the progression of dengue infection among different doses of Vitamin D and describe the dose response relationship.
4. To measure the improvement of total count of white blood cells, haematocrit and platelet count among different doses of Vitamin D and compare with the control arm to see any significance.

Study design:

Phase 2 open-label Randomized controlled trial.

Place of study:

Dengue Cell, Emergency Department and OPD of Medicine Department at Bangabandhu Sheikh Mujib Medical University (BSMMU), Shahbagh, Dhaka.

Study period:

September 2023 - August 2024 (One year)

Study population:

Potential study participants will be adults (>18 to 65years) who are NS1 positive presenting to BSMMU with fever ≥100.4°F (≥38°C) and/or typical sign symptoms of Dengue fever for 3days or less.

Sample Size:

Research instruments:

1. Structured Questionnaire
2. Check list of investigation findings

4.Centrifuge machine 5.Blood Collection set 6.RDT Kits etc.

Measures of variables:

1. Socio-Demographic variables

   1. Age
   2. Sex
   3. Residence
   4. Occupation
2. Clinical variables:

   1. Duration of fever
   2. Warning signs according to national guidelines
   3. Temperature
   4. Pulse pressure (in mm of Hg)
   5. Heart rate
   6. Respiratory rate
   7. Dengue severity grade (Group A/B/C)
3. Laboratory variables:

A. Mandatory(as a part of standard care):

1. Complete blood count - WBC, HCT, Platelet, Neutrophil:Lymphocyte ratio
2. Serum Calcium
3. Serum Albumin
4. Dengue NS1 Ag
5. Dengue IgM and IgG

B. Optional (if indicated):

* Ultrasonography of whole abdomen with lower chest

Procedure of collecting data and data analysis:

Participant enrollment and consent:

Data will be collected from the NS1 positive participants presented with fever and typical sign symptoms of dengue fever for 3days or less in Dengue cell, Emergency Department and OPD of Medicine Department in BSMMU. From the eligible participants, signed informed written consent will be obtained after explaining the purpose, procedure, potential physical and psychosocial risks, right to refuse to participate or withdraw from study. After obtaining the consent, proper history will be taken and minimum physical examination will be done and data of patient will be collected at three points in time mentioned in methodology. A detailed case record form will be prepared for data collection and used throughout the data collection period. The questionnaire will include three parts, covering demographic details, clinical information and relevant investigations.

Interventional drug information, safety and adverse effect management and recording:

The interventional drug, 2,00,000 IU Vitamin D3 oral solution in the form of cholecalciferol will be purchased from Popular pharmaceuticals LTD, which will be supplied to the patients funded by the trial. The pharmaceutical company will have no role in the trial. The drugs licence, safety and shelf life will be checked by the PI. The participants will be counselled about the potential effects of the drug. Any adverse event is very unlikely, yet will be managed by the PI and supervisor assiduously. All the adverse events will be recorded in the Case Record Form (CRF) and any drop out due to interventional effect will be reported.

Serum and plasma collection:

Following all aseptic procedure, 5 ml venous blood will be collected at enrollment day, then 4 days and 8 days thereafter. 2 ml and 3 ml will be divided in violet top and red top vacutainer respectively. The violet tube will be sent for CBC. The red tubes will be then centrifuged at 1,258 × g for 10 minutes to separate the serum and two aliquots of serum will be prepared in eppendorf tubes. One aliquot will be used to do diagnostic tests and biochemical tests. Investigations will be done from Department of Haematology, Biochemistry, Virology and Radiology of BSMMU. All investigations will be done free of cost for the patients. The remaining samples will be preserved at -80°C at study site for five years under the custody of PI and supervisors for future research purpose.

Participant's right to withdraw:

Participants are free to withdraw from study at any point, for any reason. If this occurs this reason from withdrawal will be documented in the case record form. Patients withdrawn from the study before they have undertaken study related procedures will be replaced.

Data collection, processing and analysis:

All data will be stored in an encrypted password-protected database, and the study will be conducted in accordance with Good Clinical Practice (GCP). I will be responsible to collect and record the data. The supervisor and co-supervisor will oversee the data collection. PI will be responsible for maintaining the required study records, timeliness, completeness and accuracy of the information in the Case Record Form (CRF). Data will be crosschecked by the supervisor and co-supervisor every alternate day with original source.

The numerical data obtained from the study will be entered in to excel sheet, analyzed and significance of differences will be estimated by using statistical methods and will be presented as mean ± SD or median ± IQR. Chi-square test, Mann-Whitney U-test and Kaplan-Meier curve will be done as per necessity. Different tables, graphs, charts, diagrams, etc. will be used to illustrate and publish the results of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 to 65 years.
2. NS1 positive people.
3. Fever ≥ 100.4°F (≥38°C) for 3days or less
4. Typical sign symptoms of Dengue fever.

Exclusion Criteria:

1. >72hours of fever.
2. Critically ill patients.
3. Pregnancy
4. Known Vitamin D hypersensitivity
5. High serum calcium level
6. Hypoalbuminaemia
7. Malignancy
8. Known nephrolithiasis and severe renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of mortality and progression to severe dengue. | 8 days
  Proportion of mortality and progression to severe dengue.

SECONDARY OUTCOMES:
Improvement in total count of white blood cells, haematocrit and platelet count. | 8 days
  Improvement in total count of white blood cells, haematocrit and platelet count.

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the journal authority and make public as part of the publication
Supporting Information: SAP, ICF, CSR